CLINICAL TRIAL: NCT07146750
Title: An Open-label, Phase 1, Randomized, Parallel Design Study to Determine the Bioequivalence and Investigate the Safety and Tolerability of Subcutaneous Amlitelimab Delivered by 2 Different Devices in Healthy Adult Participants
Brief Title: A Bioequivalence Study of Amlitelimab Delivered by 2 Different Devices in Healthy Adult Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEQ19340; U1111-1318-3393 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1:1:1 ratio.
Masking Description: This study is open-label. Participants, investigators, and study members have access to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): Participants will receive a single dose of subcutaneous amlitelimab (dose A) to the abdomen delivered by prefilled syringe (PFS).
  Interventions: Combination Product: SAR445229
- Group 2 (Experimental): Participants will receive a single dose subcutaneous amlitelimab (dose A) to the abdomen delivered by prefilled pen (PFP).
  Interventions: Combination Product: SAR445229
- Group 3 (Active Comparator): Participants will receive a single dose of subcutaneous amlitelimab (dose B) to the abdomen delivered by PFS.
  Interventions: Combination Product: SAR445229
- Group 4 (Experimental): Participants will receive a single dose of subcutaneous amlitelimab (dose B) to the abdomen delivered by PFP.
  Interventions: Combination Product: SAR445229

INTERVENTIONS:
Combination Product: SAR445229 — Single dose
  Other Names: Amlitelimab

SUMMARY:
This is a single-center, open-label, randomized, single-dose, parallel, Phase 1, 4-arm study designed to determine the bioequivalence and investigate the safety and tolerability profiles of subcutaneous amlitelimab delivered by 2 different devices at 2 different total doses in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female participant, between 18 and 55 years of age, inclusive, at the time of signing the informed consent form (ICF).
* Certified as healthy by a comprehensive clinical assessment [detailed medical history and complete physical examination including neurological exam (at screening and D1), skin, and mucous membranes].
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m2, inclusive.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, dermatologic, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Known history of significant immunosuppression or suspected current significant immunosuppression, including history of invasive opportunistic or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Any malignancies or history of malignancies prior to baseline (except for non-melanoma skin cancer that has been excised and cured for more than 5 years prior to baseline).
* History of solid organ (including corneal transplant) or stem cell transplant.
* Any pre-planned major elective surgery known about at baseline visit that in the Investigator's opinion would impede participation in the study.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Any nicotine use within 4 weeks before study inclusion. Regular smoking more than 5 cigarettes or equivalent in nicotine per week, unable to stop smoking or using nicotine for duration of the study.
* If female, pregnancy (defined as positive beta human chorionic gonadotropin [β-HCG] blood test), breast feeding.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
PK parameter: Cmax | From Day 1 up to End of study (approximately 24 weeks)
  Maximum serum concentration observed.
Pharmacokinetic (PK) profile: AUC last | From Day 1 up to End of study (approximately 24 weeks)
  Area under the serum concentration versus time curve calculated using the trapezoidal method from time zero to the real time.
Pharmacokinetic (PK) profile: AUC | From Day 1 up to End of study (approximately 24 weeks)
  Area under the serum concentration versus time curve extrapolated to infinity.

SECONDARY OUTCOMES:
PK parameter: Tmax | From Day 1 up to End of study (approximately 24 weeks)
  Time to reach Cmax.
PK parameter: t1/2z | From Day 1 up to End of study (approximately 24 weeks)
  Terminal half-life associated with the terminal slope (λz) determined
PK parameter: CL/F | From Day 1 up to End of study (approximately 24 weeks)
  Apparent total body clearance after a single subcutaneous administration of a drug from the serum.
PK parameter: Vz/F | From Day 1 up to End of study (approximately 24 weeks)
  Apparent volume of distribution during the terminal (λz) phase.
Pharmacokinetic (PK) profile: AUCext | From Day 1 up to End of study (approximately 24 weeks)
  Percentage of extrapolated part of AUC.
Percentage of participants who experienced TEAEs including ISRs, TESAEs, and/or TEAESIs | Up to end of study (approximately 24 weeks)
  TEAEs (Treatment-Emergent Adverse Events) including ISRs (local tolerability assessment), TESAEs (Treatment-Emergent Serious Adverse Events), and/or TEAESIs (Treatment Emergent Adverse Event of Special Interest).
Percentage of participants with potentially clinically significant abnormalities | Up to end of study (approximately 24 weeks)
  Clinically significant abnormalities including Clinical laboratory evaluations, Vital signs, electrocardiogram (ECG).
Visual analog scale score for pain with subcutaneous administration | Day 1
  VAS (visual analog scale) is used to evaluate pain at the treatment injection site. In a range between 0 to 10 where 10 is the worst pain.
Incidence of participants with ADA (antidrug antibody) against amlitelimab. | Up to end of study (approximately 24 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami- Site Number : 8400001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: BEQ19340 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26831&tenant=MT_SNY_9011